CLINICAL TRIAL: NCT02646384
Title: Ovarian Tissue Freezing For Fertility Preservation In Girls Facing A Fertility Threatening Medical Diagnosis Or Treatment Regimen
Brief Title: Ovarian Tissue Cryopreservation in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-010037
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian tissue cryopreservation (Experimental): Children faced with a fertility threatening diagnosis or treatment plan will be offered ovarian tissue cryopreservation, particularly if pre menarchal and without other options to preserve fertility. Although considered experimental, there are over 120 live births worldwide using this technique
  Interventions: Procedure: Ovarian tissue cryopreservation

INTERVENTIONS:
Procedure: Ovarian tissue cryopreservation — Ovarian tissue will be removed

SUMMARY:
The Institutional Review Board (IRB) protocol is being designed to offer ovarian tissue cryopreservation to female pediatric patients (birth-17 years of age) with fertility threatening medical diagnoses or facing surgery, chemotherapy or radiation therapy that may cause loss of reproductive potential. Because this procedure is currently considered experimental, the establishment of an IRB protocol under which this opportunity can be offered is needed.

DETAILED DESCRIPTION:
Ovarian tissue cryopreservation is currently considered experimental but offers the only opportunity for fertility preservation in pre-menarchal girls faced with a fertility threatening diagnosis or treatment plan.

ELIGIBILITY:
Inclusion Criteria: (All inclusion criteria must be met.)

1. Female, age birth-17 years
2. Meet at least one of the following three conditions:

   1. Have a diagnosis of a medical condition that is expected to result in permanent diminished or complete loss of subsequent ovarian function (e.g. Turner's syndrome) OR have a diagnosis that will create a need for surgery, chemotherapy, drug treatment and/or radiation for the treatment or prevention of the condition (e.g lupus nephritis) or malignancy and is expected to result in permanent diminished or complete loss of subsequent ovarian function. Unlike in males where a semen analysis provides an objective measure of testicular function, ovarian reserve testing remains subjective by evaluation of hormones. Therefore, to objectively qualify a degree of expected diminished loss of fertility is difficult.
   2. Or, have a medical condition or malignancy that requires removal of all or part of one or both ovaries. Girls with ovarian or germ cell tumors requiring removal of all or part of one or both ovaries will also be eligible for inclusion in the study.
   3. Or, have a newly diagnosed or recurrent disease affecting fertility.
3. For patients undergoing elective removal of all or part of an ovary for fertility preservation only, they must have two ovaries.
4. Sign an approved informed consent and authorization permitting the release of personal health information. The patient and/or the patient's legally authorized guardian must acknowledge in writing that consent for specimen collection has been obtained, in accordance with institutional policies approved by the U.S. Department of Health and Human Services.

Exclusion Criteria: (Any exclusion criteria will disqualify.)

1. Girls with psychological, psychiatric, or other conditions which prevent giving fully informed consent.
2. Girls whose underlying medical condition significantly increases their risk of complications from anesthesia and surgery.
3. Subjects with extensive disease whose therapy is deemed palliative by the medical oncologist will not be selected.
4. Subjects with suspected severe diminished ovarian reserve, such as a follicle stimulating hormone (FSH) level of > 15.

Max Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2040-01-22 (Estimated); Study Completion 2040-01-22 (Estimated)

PRIMARY OUTCOMES:
Number of pregnancy and live births after transplantation of cryopreserved ovarian tissue | 10-20 years

CONTACTS AND LOCATIONS:
Overall Officials: Zaraq Khan, M.B.B.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joshi VB, Behl S, Pittock ST, Arndt CAS, Zhao Y, Khan Z, Granberg CF, Chattha A. Establishment of a Pediatric Ovarian and Testicular Cryopreservation Program for Malignant and Non-Malignant Conditions: The Mayo Clinic Experience. J Pediatr Adolesc Gynecol. 2021 Oct;34(5):673-680. doi: 10.1016/j.jpag.2021.04.006. Epub 2021 Apr 25. PMID 33910089
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials